CLINICAL TRIAL: NCT00742937
Title: Impact of Supplementation With Dual Megadose of Vitamin A in the Post-partum About Vitamin A Levels in Breast Milk, Serum Levels of Vitamin A and Iron in the Binomial Mother-son and Growth and Morbidity of Children Under 6 Months
Brief Title: Impact of Maternal Supplementation With Dual Megadose of Vitamin A
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Ilma Kruse Grande de Arruda, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMIPVITA-001
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Hypovitaminosis; Vitamin A Deficiency
Keywords: Hypovitaminosis A
MeSH Terms: conditions — Avitaminosis; Vitamin A Deficiency | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): After birth the women will receive one capsule 200,000 UI of retinol palmitate (vitamin A)plus vitamin E and eight days after delivery the second capsule of vitamin E will be administer.
  Interventions: Dietary Supplement: Placebo
- B (Experimental): After birth the women will receive one capsule 200,000 UI of retinol palmitate (vitamin A)plus vitamin E and eight days after delivery the second capsule of 200,000 UI of retinol palmitate (vitamin A)plus vitamin E will be administer.
  Interventions: Dietary Supplement: vitamin A

INTERVENTIONS:
Dietary Supplement: vitamin A — second capsule 200,000 UI of retinol palmitate (vitamin A)plus vitamin E, eight days after delivery.
  Arms: B
Dietary Supplement: Placebo — second capsule with vitamin E, eight days after delivery.
  Arms: A

SUMMARY:
The purpose of this study is to evaluate the effect of maternal supplementation with 400,000 IU of oral retinol palmitate in the post-partum, the nutritional situation of the binomial mother-child, on growth and morbidity of children in breastfeeding in the first six months of life.

DETAILED DESCRIPTION:
The effect will be assessed by the milk and blood.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant low-risk obstetric

Exclusion Criteria:

* Premature birth
* Newborn babies with birth defects and / or other serious diseases

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Seric retinol | six months

SECONDARY OUTCOMES:
Morbidity and growth of the child. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Ilma Kruze, PhD, Principal Investigator
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Tomiya MT, de Arruda IK, da Silva Diniz A, Santana RA, da Silveira KC, Andreto LM. The effect of vitamin A supplementation with 400 000 IU vs 200 000 IU on retinol concentrations in the breast milk: A randomized clinical trial. Clin Nutr. 2017 Feb;36(1):100-106. doi: 10.1016/j.clnu.2015.11.018. Epub 2015 Dec 17. PMID 26725194
- [Derived] Dos Santos CS, Kruze I, Fernandes T, Andreto LM, Figueiroa JN, Diniz Ada S. The Effect of a Maternal Double Megadose of Vitamin A Supplement on Serum Levels of Retinol in Children Aged under Six Months. J Nutr Metab. 2013;2013:876308. doi: 10.1155/2013/876308. Epub 2013 Dec 24. PMID 24455219
- [Derived] Fernandes TF, Figueiroa JN, Grande de Arruda IK, Diniz Ada S. Effect on infant illness of maternal supplementation with 400 000 IU vs 200 000 IU of vitamin A. Pediatrics. 2012 Apr;129(4):e960-6. doi: 10.1542/peds.2011-0119. Epub 2012 Mar 12. PMID 22412025